CLINICAL TRIAL: NCT03502642
Title: Ropivacaine Continuous Wound Infusion Versus Intrathecal Morphine for Postoperative Analgesia After Cesarean Delivery : A Randomized Controlled Trial
Brief Title: Ropivacaine Continuous Wound Infusion Versus Intrathecal Morphine for Postoperative Analgesia After Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Collaborators: LEVENTON (Unknown)
Responsible Party: Principal Investigator, Hicham Abou Zeid, Assistant Professor, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEHDF944
Record Dates: First submitted 2018-03-23; First posted 2018-04-19 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Obstetric Pain
Keywords: Ropivacaine; wound infusion; analgesia; cesarean; intrathecal morphine; randomized controlled trial
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Anesthesia, Spinal; Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: healthy, term women scheduled for cesarean delievry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (P) (Placebo Comparator): Placebo group parturients will receive spinal anesthesia with intrathecal morphine and will have continuous normal saline wound infusion (Dosi-Pain® Kit, LEVENTON SAU, Spain).
  Interventions: Device: wound infusion (Dosi-Pain® Kit, LEVENTON SAU, Spain); Procedure: Spinal Anesthesia; Drug: intrathecal morphine; Drug: Normal saline
- Ropivacaine (R) (Active Comparator): Ropivacaine group parturients will receive spinal anesthesia without intrathecal morphine and will have continuous ropivacaine (Ropivacaina Molteni®) wound infusion (Dosi-Pain® Kit, LEVENTON SAU, Spain).
  Interventions: Device: wound infusion (Dosi-Pain® Kit, LEVENTON SAU, Spain); Procedure: Spinal Anesthesia; Drug: Ropivacaine (Ropivacaina Molteni®)

INTERVENTIONS:
Device: wound infusion (Dosi-Pain® Kit, LEVENTON SAU, Spain) — After peritoneum closure a 16cm multiorifice perforated catheter (Dosi-Pain® Kit, LEVENTON SAU, Spain) was inserted by the surgeon below the fascia used for normal saline continuous infusion in the Placebo group and for continuous ropivacaine infusion (Ropivacaina Molteni®, MOLTENI FARMACEUTICI, Italy) in the ropivacaine group.
  Other Names: wound catheter
Procedure: Spinal Anesthesia — Cesarean section was conducted under spinal anesthesia in both groups
Drug: intrathecal morphine — Intrathecal morphine was administered during spinal anesthesia in the placebo group but not in the ropivacaine group
  Arms: Placebo (P)
Drug: Ropivacaine (Ropivacaina Molteni®) — A10ml bolus of ropivacaine 7.5mg/ml were administered in the wound catheter after skin closure then an infusion of ropivacaine 2mg/ml at the rate of 5ml/h was administered as wound infusion via the Dosi-Pain® Kit for 48hours.
  Arms: Ropivacaine (R)
Drug: Normal saline — A10ml bolus of normal saline were administered in the wound catheter after skin closure then an infusion of normal saline at the rate of 5ml/h was administered as wound infusion via the Dosi-Pain® Kit for 48hours.
  Other Names: Placebo
  Arms: Placebo (P)

SUMMARY:
Cesarean delivery is one of the most common surgical procedures, performed at an increasingly high rate. It is associated with intense postoperative pain that may hamper the rehabilitation process and interfere with patient satisfaction and care provided to the newborn. Therefore, control of perioperative pain with multimodal regimens using local anesthetic may be important in short- and long-term convalescence after surgery.

Opioid-based regimens are the "gold standard" of cesarean delivery analgesia. However, spinal and epidural opioids have a ceiling effect.

Wound infiltration with local anesthetics has been used widely in the multimodal approach of pain relief. Continuous wound infusion with local anesthetic through a multiorifice catheter increases the duration of action and efficacy of local surgical wound infiltration compared with a one-time wound injection of local anesthetic.

After cesarean delivery, Local anesthetic continuous wound infusion would be associated with better reduction in pain scores when compared to intrathecal morphine . Therefore, an assessor and patient blinded, randomized study that aimed to compare the efficacy and side effects of these analgesia techniques was conducted.

ELIGIBILITY:
Inclusion Criteria:

* women.
* age between 18 and 50 years.
* gestational age 37 to 42 weeks.
* body mass index ranging from 18.0 to 30.0 kg/m2
* American Society of Anesthesiology (ASA) physical status I or II
* elective cesarean delivery with a Pfannenstiel incision
* spinal anesthesia.

Exclusion Criteria:

* history of chronic opioid use.
* Allergy to opioids and or local anesthetics.
* absolute or relative contraindication to neuraxial anesthesia.
* fever or any other sign of infection.
* Diabetes Mellitus under insulin therapy
* physical separation of patients from the neonate during the postoperative period.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
pain at rest | Hour 0, Hour 2, Hour 6, Hour 12, Hour 24, Hour 36 and Hour 48
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at rest | Hour 2
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at rest | Hour 6
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain.Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at rest | Hour 12
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain.Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at rest | Hour 24
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain.Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at rest | Hour 36
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at rest | Hour 48
  Pain scores at rest were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain.Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.

SECONDARY OUTCOMES:
pain at mobilization | Hour 0
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at mobilization | Hour 2
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at mobilization | Hour 6
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at mobilization | Hour 12
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at mobilization | Hour 24
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at mobilization | Hour 36
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
pain at mobilization | Hour 48
  Pain scores at mobilization were measured postoperatively using visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain. Measures were repeated for 48hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 0
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 2
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 6
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 12
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 24
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 36
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of postoperative nausea and vomiting | Hour 48
  incidence of postoperative nausea and vomiting. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 0
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 2
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 6
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 12
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 24
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 36
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of pruritus | Hour 48
  incidence of pruritus. Measurements were made for 48 hours postoperatively.Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of urinary retention | during the 48 hours postoperatively
  defined as the requirement of bladder recatheterization postoperatively.
return of gastrointestinal function | during the 48 hours postoperatively
  interval from the end of surgery until first gas elimination postoperatively. interval from the end of surgery until first feces elimination postoperatively.
sedation | Hour 0
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
sedation | Hour 2
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
sedation | Hour 6
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
sedation | Hour 12
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
sedation | Hour 24
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
sedation | Hour 36
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
sedation | Hour 48
  assessed by a 5-point rating scale (0 fully alert,
  1 sleepy but easily aroused with verbal stimulation, 2 sleepy but aroused with light touch, 3 sleepy but aroused with pain, and 4 unconscious patient). Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 0
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 2
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 6
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 12
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 24
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 36
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.
incidence of neurological alterations | Hour 48
  patients were specifically asked about paresthesia, tactile hyperesthesia, and headache. Measurements were made for 48 hours postoperatively. Hour 0 is the time of arrival to the post anesthesia care unit PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Hicham A Abou Zeid, M.D., Study Chair — Saint Joseph University- Lebanon; Nicole M Naccahe, M.D., Study Director — Saint Joseph University- Lebanon; Samer H Hotayt, M.D., Principal Investigator — Saint Joseph University- Lebanon
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No